CLINICAL TRIAL: NCT00991055
Title: To Compare the Efficacy and Safety Between Pioglitazone Added to Combination Therapy of Sulfonylurea Plus Metformin and Placebo Control Group in Patients With Type 2 Diabetes
Brief Title: Comparison of the Efficacy and Safety Between Pioglitazone and Placebo Added to Combination Therapy in Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: National Cheng-Kung University Hospital, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HR-96-61
Record Dates: First submitted 2009-10-01; First posted 2009-10-07 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone (Experimental)
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator)
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — A total 16-week randomized, double-blind, controlled study to compare the efficacy and safety of pioglitazone 15mg once daily added to combination metformin plus sulfonylurea with those of placebo combining control group.
  (4-week run in period and 12-week pioglitazone 15mg added to combination therapy of sulfonylurea plus metformin and placebo control group in patients with type 2 diabetes)

SUMMARY:
The purpose of this trial is to study the efficacy and safety of pioglitazone added to combination therapy of sulfonylurea plus metformin with placebo in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Pioglitazone hydrochloride, a thiazolidinedione compound, is a new therapeutic agent for the treatment of type 2 diabetes that reduces insulin resistance by enhancing insulin action in skeletal muscle, liver, and adipose tissue. In the study of diabetes, pioglitazone reduced the hyperglycemia, hyperinsulinemia, and hypertriglyceridemia characteristic of insulin-resistant states. The metabolic changes induced by pioglitazone result in increased responsiveness of insulin-dependent tissues and are observed in numerous models of insulin resistance.

In the present randomized, double-blind, parallel study, we aim to compare the efficacy and safety of pioglitazone added to combination therapy of sulfonylurea plus metformin with those of sulfonylurea plus metformin for the treatment of type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, Aged > 25 years and had been diagnosed as type 2 diabetes for at least 3 months before study entry.
2. Subjects have taken sulfonylurea plus metformin therapy for at least 3 months before study entry.
3. Subjects have to take daily Metformin 500~2000mg tolerable dosages and sulfonylurea (such as the usage dose of glimepiride ≧4mg; dose of Gliclazide≧160mg; dose of Glipizide ≧20mg; dose of glyburide≧4mg) for at least 1 months.
4. Those subjects with HbA1C historical levels between 7.0% and 11.0% within 3 month prior to study entry.
5. BMI between 20-35 kg /m2.
6. Each subject must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document.
7. Subjects have been under stable diet control for at least 1 month before study entry.
8. Subjects are willing to stick to current diet and sulfonylurea plus metformin treatment plan during this trial.

Exclusion Criteria:

1. Pregnant women or lactating mothers.
2. Type 1 DM(IDDM), or diabetes caused by pancreas damage、secondary forms of diabetes, i.e., Cushing's syndrome or acromegaly.
3. A history of acute metabolic complication within 3 months before study entry, i.e., ketoacidosis or hyperosmolar state (coma).
4. There are significant macrovascular complications (i.e. unstable angina or acute myocardial infarction) or renal impairment (serum creatinine higher than 1.5 mg/dL).
5. Have a known allergy to pioglitazone.
6. Other medications can be taken if their use had been instituted before study entry, but agents that can interfere with study evaluations, including other oral antidiabetic agents and corticosteroids, were not allowed.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-06 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in HbA1Cand FPG | Week 12

SECONDARY OUTCOMES:
Insulin resistance (HOMA-IR index) | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Ta-Jen Wu, MD, Principal Investigator — National Cheng Kung University College and Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan